CLINICAL TRIAL: NCT00311025
Title: Stroke: Reduction of Physical Performance Post Stroke. Inactivity or Secondary Complications? How to Cope Daily Life Activities for as Long as Possible.
Brief Title: Stroke: Reduction of Physical Performance Post Stroke. Inactivity or Secondary Complications?
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Oslo University College (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Educational/Counseling/Training
Other Study IDs: S-03054
Record Dates: First submitted 2006-04-03; First posted 2006-04-05 (Estimated); Last update posted 2006-04-05 (Estimated); Status verified 2005-09

CONDITIONS: Cerebral Stroke
Keywords: stroke; physical therapy; rehabilitation; exercise; longterm follow-up
MeSH Terms: conditions — Stroke; Motor Activity

INTERVENTIONS:
Procedure: intensive endurance, strength and balance exercises

SUMMARY:
The purpose of this project is to follow first-ever- acute stroke patients from onset, one, two and four years post stroke and study the effect of two different approaches of exercises implemented the first year post-stroke.

DETAILED DESCRIPTION:
Stroke is a major cause of disability and the long-term effects of stroke often lead to need of rehabilitation services. It has been shown that intensive stroke unit care and functional exercises are beneficial in the acute rehabilitation of stroke. The duration of the rehabilitation of patients with acute stroke is decreasing, leaving patients with not complete recovery at discharge in need of follow-up services. There is a general assumption that physical exercises are beneficial at all stages of stroke but it is questionable if these benefits are sustained after treatment ends. There are, to our knowledge, no longitudinal studies of non-interrupted regular physical exercises from the acute phase till one year post stroke.

The purpose of this project is to follow first-ever- acute stroke patients from onset, one, two and four years post stroke. All acute stroke patients will be treated in a stroke unit and the physiotherapy treatment will be according to Motor Relearning Programme principles with functional goals, environmental context and early mobilisation. When patients are discharged they will be block randomised and stratified according to gender and hemisphere lesion into two groups. Group 1 will be offered an intensive follow-up programme, which will run four times in the post-stroke year with a total amount of 80 hours of physiotherapy. The physiotherapy treatment will be focused on physical endurance, strength and balance.

Group 2, or the control group, will be offered the same physiotherapy programme that is practised within the community as of now (2003) that is when the need for follow-up is considered by someone involved. The physiotherapy then given is according to specified needs e.g. walking capacity, transfers and assistive devices.

ELIGIBILITY:
Inclusion Criteria:

* First-time ever stroke
* Neurological signs
* Computer tomography confirmed stroke
* Voluntary participation

Exclusion Criteria:

* Subarachnoid bleeding
* Tumour
* Other serious illness
* Brain stem or cerebellum stroke

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60
Dates: Start 2003-09; Study Completion 2005-09

PRIMARY OUTCOMES:
Motor Assessment Scale

SECONDARY OUTCOMES:
Bergs Balance Scale,
Timed-Up-and-Go,
6 minute walk test,
Nottingham Health Profile,
Martin Vigorimeter,
Ashworth Scale,
Barthel ADL index,
Fillenbaum´s I-ADL,
blood pressure,
heart rate

CONTACTS AND LOCATIONS:
Overall Officials: Birgitta M Langhammer, phd student, Principal Investigator — Oslo University College
Locations (1):
- Sykehuset Asker og Bærum HF, Postboks 83,, Rud, Norway